CLINICAL TRIAL: NCT02884843
Title: A Comparative Randomized Prospective Study Between the New Intubating Laryngeal Tube Suction-Disposable and the Ambu AuraGain in Blind and Fibreoptic-guided Intubation
Brief Title: The New Intubating Laryngeal Tube Suction-Disposable
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, Medical Doctor, Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: BnaiZionMC-16-LG-004
Record Dates: First submitted 2016-08-15; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Laryngeal Tube; blind intubation; fiberoptic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation laryngeal Tube Suction (Active Comparator): Intubation laryngeal Tube Suction Disposable
  Interventions: Device: Intubation laryngeal Tube Suction
- AuraGain Laryngeal Mask (Active Comparator): AuraGain Laryngeal Mask
  Interventions: Device: AuraGain Laryngeal Mask

INTERVENTIONS:
Device: Intubation laryngeal Tube Suction — Intubation laryngeal Tube Suction
  Arms: Intubation laryngeal Tube Suction
Device: AuraGain Laryngeal Mask — AuraGain Laryngeal Mask
  Arms: AuraGain Laryngeal Mask

SUMMARY:
The study compares the intubating Laryngeal Tube Suction (iLTS-D) with the Ambu®AuraGain™ in blind and fibreoptic endotracheal intubation.

The current randomized study is designed to assess the success rate of blind and fibreoptic endotracheal intubation using i-LTS-D, in comparison with the Air-Q, i-gel® and Ambu®AuraGain™ in an airway simulator. The investigators hypothesize that the iLTS-D and the Supreme Laryngeal Mask Airway will similarly perform during spontaneous ventilation despite differences in their structural design.

DETAILED DESCRIPTION:
The intubating Laryngeal Tube Suction-Disposable (iLTS-D) (VBM Medizintechnik, Sulz, Germany) is a new updated version of the Laryngeal Tube-Suction Disposable (LTS-D).

It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube (ETT) either blindly or with fibreoptic guidance. Similarly to the LTS-D, the iLTS-D also has a separate channel for gastric tubes placement up to a size of 18 Fr.

The current randomized study was designed to assess the success rate of blind and fibreoptic endotracheal intubation using iLTS-D, in comparison with the Ambu® AuraGain™ in adult patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology I and II

Exclusion Criteria:

* Difficult intubation, cervical pathology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time of blind intubation measure in seconds | 30 seconds

SECONDARY OUTCOMES:
Time of Fiberoptic intubation measure in seconds | 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Luis a Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes